CLINICAL TRIAL: NCT04210752
Title: A Phase 1, Randomised, Activator-Controlled, Double-Blind, Parallel Study to Assess the Safety, Tolerability and Explore the Immunogenicity of EG-HZ in Healthy Adult Volunteers
Brief Title: Study to Assess the Safety, Tolerability and Explore the Immunogenicity of EG-HZ in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EyeGene Inc. (Other)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EG-HZ-101
Record Dates: First submitted 2019-12-17; First posted 2019-12-26 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Prevention of Herpes Zoster (HZ)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment 1 (EG-HZ-001) (Experimental): Subjects will receive two single IM vaccinations, 2 months apart, the first on Day 1 and the second on Day 60 (±5 days). Subjects will be randomised to treatment at a ratio of 1:1:1:1:1 (n=8 per treatment)
  Route of administration: Intramuscular injection
  Interventions: Drug: Treatment 1 (EG-HZ-001)
- Treatment 2 (EG-HZ-002) (Experimental): Subjects will receive two single IM vaccinations, 2 months apart, the first on Day 1 and the second on Day 60 (±5 days). Subjects will be randomised to treatment at a ratio of 1:1:1:1:1 (n=8 per treatment)
  Route of administration: Intramuscular injection
  Interventions: Drug: Treatment 2 (EG-HZ-002)
- Treatment 3 (EG-HZ-003) (Experimental): Subjects will receive two single IM vaccinations, 2 months apart, the first on Day 1 and the second on Day 60 (±5 days). Subjects will be randomised to treatment at a ratio of 1:1:1:1:1 (n=8 per treatment)
  Route of administration: Intramuscular injection
  Interventions: Drug: Treatment 3 (EG-HZ-003)
- Treatment 4 (EG-HZ-004) (Experimental): Subjects will receive two single IM vaccinations, 2 months apart, the first on Day 1 and the second on Day 60 (±5 days). Subjects will be randomised to treatment at a ratio of 1:1:1:1:1 (n=8 per treatment)
  Route of administration: Intramuscular injection
  Interventions: Drug: Treatment 4 (EG-HZ-004)
- Treatment 5 (Shingrix) (Experimental): Shingrix
  Suspension for injection supplied as a single dose vial of lyophilised VZVgE antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. After reconstitution, a single dose of ShingrixTM is 0.5 mL.
  Route of Administration: Intramuscular injection
  Interventions: Drug: Treatment 5

INTERVENTIONS:
Drug: Treatment 1 (EG-HZ-001) — Subjects will receive two single IM vaccinations, 2 months apart, the first on Day 1 and the second on Day 60 (±5 days). Subjects will be randomised to treatment at a ratio of 1:1:1:1:1 (n=8 per treatment)
  Route of Administration: IM injection
  Other Names: EG-HZ
  Arms: Treatment 1 (EG-HZ-001)
Drug: Treatment 2 (EG-HZ-002) — Subjects will receive two single IM vaccinations, 2 months apart, the first on Day 1 and the second on Day 60 (±5 days). Subjects will be randomised to treatment at a ratio of 1:1:1:1:1 (n=8 per treatment)
  Route of Administration: IM injection
  Other Names: EG-HZ
  Arms: Treatment 2 (EG-HZ-002)
Drug: Treatment 3 (EG-HZ-003) — Subjects will receive two single IM vaccinations, 2 months apart, the first on Day 1 and the second on Day 60 (±5 days). Subjects will be randomised to treatment at a ratio of 1:1:1:1:1 (n=8 per treatment)
  Route of Administration: IM injection
  Other Names: EG-HZ
  Arms: Treatment 3 (EG-HZ-003)
Drug: Treatment 4 (EG-HZ-004) — Subjects will receive two single IM vaccinations, 2 months apart, the first on Day 1 and the second on Day 60 (±5 days). Subjects will be randomised to treatment at a ratio of 1:1:1:1:1 (n=8 per treatment)
  Route of Administration: IM injection
  Other Names: EG-HZ
  Arms: Treatment 4 (EG-HZ-004)
Drug: Treatment 5 — Shingrix
  Suspension for injection supplied as a single dose vial of lyophilised VZVgE antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. After reconstitution, a single dose of ShingrixTM is 0.5 mL.
  Route of Administration: IM injection
  Other Names: Comparator
  Arms: Treatment 5 (Shingrix)

SUMMARY:
This is a Phase 1, first in human (FIH), randomised, active-controlled, double-blind study designed to assess the safety and tolerability and explore preliminary efficacy of the EG-HZ vaccine. Oversight will be provided by a Safety Review Committee (SRC).

DETAILED DESCRIPTION:
Subjects will undergo a Screening period beginning up to 28 days prior to randomisation, the first of two vaccinations administered 2 months apart, pre- and post-dose assessment, follow-up visits, and an end of study (EOS) or early termination (ET) visit (as applicable).

Subjects will be randomised prior to vaccination on Day 1, to one (1) of five (5) treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent before the first study-specific procedure;
2. Healthy male and female volunteers aged 50 to 70 years at time of Screening;
3. Subjects must have a BMI between ≥18.0 and ≤35.0 kg/m2 at Screening;
4. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements;
5. Must have a negative urine pregnancy test on the day of dosing prior to each vaccination;
6. Subjects must have clinical laboratory values within normal ranges as specified by the testing laboratory, unless deemed NCS by the PI;
7. Normal physical findings, vital signs, 12-lead ECG, and no significant medical condition at the time of Screening, as judged by the PI;
8. Must agree to abstain from alcohol intake from 48 hours before each vaccination;
9. Must be non-smokers or, if light or occasional smokers (<10 cigarettes per day), must agree to abstain from smoking from 48 hours before each vaccination;
10. Must have a negative urine drug screen/alcohol breath test on the day of dosing prior to each vaccination. Repeat urine drug screens will be permitted for suspected false positive results;
11. Must agree to use highly effective, medically accepted double-barrier contraception (both male and female partners) from Screening until study completion as specified below in this criterion. Highly effective double-barrier contraception is defined as use of a condom

AND one of the following:

1. Birth control pills (The Pill)
2. Depot or injectable birth control
3. IUD
4. Birth Control Patch (e.g., Ortho Evra)
5. NuvaRing®
6. Implantable contraception (e.g., Implanon)
7. Documented evidence of surgical sterilisation at least 6 months prior to Screening, i.e., tubal ligation or hysterectomy for women or vasectomy for men

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period;
2. History of severe allergic reaction (e.g., anaphylaxis) to any component of the vaccine;
3. History of herpes zoster (Shingles);
4. Previous vaccination against HZ (either a registered product or an investigational product through participation in a HZ vaccine study);
5. Previous vaccination against VZV;
6. Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within 3 months prior to the first vaccine dose (intra-articular, intra-bursal, or topical [skin or eyes] corticosteroids are permitted at the discretion of the PI);
7. History of autoimmune disease/s which required therapeutic intervention/s, or any active autoimmune disease requiring therapeutic intervention/s including but not limited to: systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenic purpura, glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and insulin-dependent diabetes mellitus (i.e. type 1 diabetes);
8. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the Investigator, contraindicate intramuscular injection;
9. Vaccines administered or scheduled in the period from 4 weeks prior to Dose 1 through to 28 days post-vaccination dose 2, excluding licensed non-replicating vaccines (i.e., inactivated and subunit vaccines, including inactivated and subunit influenza vaccines for seasonal or pandemic flu, with or without adjuvant) administered up to 8 days prior to each dose and/or at least 14 days after any dose of study vaccine (to be determined at the discretion of the PI);
10. Receipt of any immunoglobulins or blood/plasma products within 60 days prior to vaccination on Day 1 and until the EOS/ET visit;
11. Positive test for HCV, HBsAg, or HIV antibody at Screening;
12. History or presence of any clinically unstable medical, surgical or psychiatric condition, at the discretion of the Investigator;
13. Active malignancy and/or history of malignancy in the past 5 years, except for completely excised basal cell carcinoma or low grade cervical intraepithelial neoplasia;
14. History of significant hypersensitivity or anaphylaxis involving any drug, food or other precipitating agent (e.g., bee sting);
15. Abnormal laboratory values or investigations (including ECG) that, in the opinion of the Investigator, are deemed clinically significant and would preclude participation in the study;
16. Renal insufficiency defined by eGFR <90 mL/min (CKD-EPI);
17. Hepatic synthetic insufficiency as defined as a serum albumin of <35 g/L; or serum bilirubin >20 μmol/L;
18. Acute disease or acute stage of chronic disease and/or fever at the time of enrolment. Fever is defined as temperature ≥ 37.5°C (99.5°F), regardless of the route. Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the Investigator;
19. Regular use of any prescribed or non-prescribed medications, including herbal remedies, which, in the opinion of the Investigator, might adversely affect the safety of the subject or the interpretability of study results. Participants who are taking a stable dose of medication for a controlled medications include, for example, stable doses of antidepressants, cholesterol lowering agents, high blood pressure medication, reflux medication, hormone replacement therapy, NSAIDs, paracetamol, occasional Ventolin, etc.);
20. History of or present alcohol abuse, or excessive intake of alcohol, as judged by the Investigator;
21. Blood donation or significant blood loss within 30 days prior to the first study drug administration and until the EOS/ET visit;
22. Plasma donation within 7 days prior to the first study drug administration and until the EOS/ET visit;
23. Administration of another IP (defined as a compound that has not been approved for marketing) or has participated in any other clinical study that included IP treatment within 3 months prior to administration of IP in this study;
24. Any person who is initially excluded from study participation based on one or more of the time-limited exclusion criteria (e.g., acute illness) may be considered for enrollment once the condition has resolved as long as the subject continues to meet all other entry criteria;
25. Subject taking any non-topical antiviral therapy with activity against herpes viruses, including but not limited to acyclovir, famciclovir, ganciclovir, and valacyclovir 3 days prior to vaccination or 14 days after;
26. Any other reason that, in the opinion of the Investigator, might interfere with the evaluation required by the study;
27. The subject is, in the opinion of the Investigator, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, estimated 9 months
  Safety and tolerability determined by abnormal clinical laboratory tests, vitals signs, physical exam, ECG parameters. It is an composite Outcome

SECONDARY OUTCOMES:
To explore the immunogenicity of EG-HZ at various excipient combinations | Blood samples for analysis of immunogenicity will be collected pre-dose and at multiple time points post-dose following administration of each vaccination. Through study completion, estimated 9 months
  Immunogenicity is determined by Anti-Glycoprotein E total immunoglobulin G (IgG) antibody concentration at 1 month (Day 90) and 6 months (Day 240) post last vaccination.
  Humoral immunity: anti-Varicella zoster virus total IgG antibody; anti-Glycoprotein E total IgG antibody.
  Cell-mediated immunity: CD4+ T cell; CD8+ T cell

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Ltd (Nucleus Network), Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954